CLINICAL TRIAL: NCT00876434
Title: Subconjunctival Sirolimus for the Treatment of Autoimmune Active Anterior Uveitis
Brief Title: Subconjunctival Sirolimus for the Treatment of Autoimmune Active Anterior Uveiti
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090116; 09-EI-0116
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-02-10

CONDITIONS: Anterior Uveitis
Keywords: Sirolimus; Anterior Uveitis; Autoimmune Disease; Uveitis
MeSH Terms: conditions — Uveitis, Anterior; Autoimmune Diseases; Uveitis | interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus

SUMMARY:
Background:

* Uveitis is an inflammatory condition in which the patient's own immune system attacks the eye, causing eye inflammation and vision loss. Patients with uveitis may be treated with immunosuppressive medications to reduce the inflammation and prevent vision loss.
* Sirolimus is an immunosuppressive medication that is approved by the U.S. Food and Drug Administration (FDA) to prevent organ rejection following a kidney transplant. Researchers think that sirolimus may affect the part of the immune system that may be an important cause of uveitis, and may decrease the inflammation that causes uveitis.
* In this study, sirolimus will be given as an injection under the outer layer of your eye. The FDA has permitted the investigational use of sirolimus for this study.

Objectives:

* To determine if subconjunctival injection of sirolimus is safe for treatment of uveitis.
* To see if sirolimus is an effective treatment for uveitis.

Eligibility:

* Patients 18 years of age and older with active uveitis in one or both eyes. If a patient has uveitis in both eyes, the one in which the inflammation is worse will be treated during the study. The vision in the study eye must be at least 20/400.
* Patients must have good liver function, and must be willing to practice sun protection measures for 2 weeks following the treatment.

Design:

* Treatment with sirolimus in the study eye:
* Antibiotic and numbing eye drops will be given before the sirolimus injection.
* 1 dose of sirolimus will be injected directly into the subconjunctiva (white part of the eye).
* Antibiotic drops will be given for topical application 3 times per day for 2 days after the injection.
* Patients will be followed for 16 weeks after sirolimus injection (initial visit and follow-up visits in Weeks 2, 4, 8, 12, and 16).
* Evaluations during the treatment period and follow-up visits:
* Physical examination, including vital signs and body weight checks, and pregnancy test for women who can become pregnant.
* Full medical and ophthalmic history, involving questionnaires and discussion with researchers.
* Eye examination, dilation, and photography, including measurements of retinal thickness and fluorescent dye tests of blood flow in the eye.
* Blood and urine tests.
* Because of the increased risk of skin cancer associated with sirolimus, patients ...

DETAILED DESCRIPTION:
Objective: Uveitis refers to intraocular inflammatory diseases that are an important cause of visual loss. Standard systemic immunosuppressive medications for uveitis can cause significant adverse effects and many patients continue to experience disease flare-ups. Sirolimus suppresses cytokine-driven T-cell proliferation and thus, inhibits the production, signaling and activity of many growth factors relevant to uveitis. Subconjunctival sirolimus administration could reduce or eliminate the need for topical and/or systemic immunosuppressive drugs that could result in reduced morbidity. This protocol will investigate subconjunctival sirolimus as a possible treatment for active anterior uveitis.

Study Population: Five participants with active anterior uveitis will be initially accrued in this study. Participants must require treatment for their uveitis with systemic and/or topical anti-inflammatory medications at high frequency intervals [greater than or equal to three times daily (T.I.D.)] or local steroid treatment (periocular steroid injections) is contraindicated because of significant intraocular pressure (IOP) elevation with local steroid treatments in the past (i.e., steroid responder), have at least a grade of 1+ for anterior chamber cells and have visual acuity of at least 20/400 in the study eye. Up to seven participants may be enrolled, as up to two participants may be accrued to replace enrolled participants who withdraw from the study prior to receiving any study medication.

Design: This is a Phase I, non-randomized, prospective, uncontrolled single-center study to evaluate subconjunctival sirolimus as a treatment for active anterior uveitis. All participants will receive a single 30-microL (1,320 microg) subconjunctival sirolimus injection in the study eye at baseline and will be followed for 16 weeks post-injection.

Outcome Measures: The primary outcome is the number of participants who experience at least a 2-step reduction in anterior chamber inflammation within four weeks post-injection. Secondary outcomes include changes in visual acuity and anterior chamber inflammation grading, the number of participants who experience a disease flare within the 16-week study duration and, of the participants who experience a disease flare, the number of days to disease flare from baseline. Secondary outcomes also include the presence or extent of cystoid macular edema.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participant has the ability to understand and sign the informed consent document.
* Participant is 18 years of age or older.
* Participant's uveitis is considered active on current regimen.
* Participant has a diagnosis of non-infectious anterior uveitis requiring treatment to control their intraocular inflammatory disease with systemic and/or topical anti-inflammatory medications at high frequency intervals (greater than or equal to T.I.D.) or local steroid treatment (periocular steroid injections) is contraindicated because of significant IOP elevation with local steroid treatments in the past (steroid responder).
* Participant has anterior uveitis with at least a grade of 1+ for anterior chamber cells 1 in the study eye.
* Participant has visual acuity in the study eye of 20/400 or better (or ETDRS equivalent).
* Participant has normal renal or liver function, or no worse than mild abnormalities as defined by the Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
* Participant has no history of intraocular surgery within three months prior to study enrollment and agrees not to undergo elective ocular surgery (e.g., cataract extraction) for the duration of the study.
* Participant has an absolute neutrophil count (ANC) above 750/mm(3)
* Participant is able to undergo full ophthalmic examination for assessment of anterior chamber cells.
* Participant understands there is an increased risk for skin cancer with sirolimus usage and agrees to practice skin protective measures for two weeks following their injection. Skin protective measures include: 1) staying out of direct sunlight, especially between the hours of 10:00 a.m. and 3:00 p.m., if possible; 2) wearing protective clothing, including a hat and sunglasses; 3) applying a sun block product that has a skin protection factor (SPF) of at least 15 (some participants may require a product with a higher SPF number, especially if they have a fair complexion); 4) applying a sun block lipstick that has a SPF of at least 15 to protect the lips; and 5) not using a sun lamp or tanning booth or bed.
* Participant is willing and able to comply with the study procedures.
* Female participants of childbearing potential must not be pregnant or breast-feeding, must have a negative urine pregnancy test at screening and must be willing to undergo urine pregnancy tests throughout the study.
* Both female participants of childbearing potential and male participants able to father a child must agree to practice two forms of adequate birth control throughout the course of the study and for three months post-injection. Acceptable methods of birth control include hormonal contraception (birth control pills, injected hormones or vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom and spermicide) or surgical sterilization (hysterectomy, tubal ligation or vasectomy).

  * Participants with a hysterectomy or vasectomy (or have a partner with a hysterectomy or vasectomy) are exempt from using two methods of contraception. However, female participants with a tubal ligation (or male participants who have a female partner with a tubal ligation) are not exempt, and are required to practice another acceptable method of birth control.

EXCLUSION CRITERIA:

* Participant has a significant active infection (an infection requiring treatment as determined by the medical team) or a history of chronic or recurrent infections.
* Participant has a history of cancer (other than a non-melanoma skin cancer) diagnosed within the past five years.
* Participant has used latanoprost (Xalatan (Registered Trademark)) within two weeks prior to study enrollment or is likely to need it at any point during the study as determined by the investigator.
* For participants with active anterior uveitis in both eyes, the participant's non-study eye is anticipated to require periocular steroids or it is anticipated that an increase in systemic immunosuppressive treatments including steroids may be required during the course of the study.
* Participant has a media opacity that precludes assessment of anterior chamber inflammation.
* Participant has active joint or systemic inflammation requiring immediate addition or increase in systemic anti-inflammatory medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-04-01; Primary Completion 2011-02-10 (Actual); Study Completion 2011-02-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the number of participants who experience at least a 2-step reduction in inflammation within four weeks post-injection.

SECONDARY OUTCOMES:
Changes in VA; changes in AC cells & flare-ups; number of disease flares, number of days until the first disease flare; the presence or extent of CME; the amount of retino-vascular leakage; and changes in retinal thickening.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117
- [Background] Gritz DC, Wong IG. Incidence and prevalence of uveitis in Northern California; the Northern California Epidemiology of Uveitis Study. Ophthalmology. 2004 Mar;111(3):491-500; discussion 500. doi: 10.1016/j.ophtha.2003.06.014. PMID 15019324
- [Background] Wakefield D, Dunlop I, McCluskey PJ, Penny R. Uveitis: aetiology and disease associations in an Australian population. Aust N Z J Ophthalmol. 1986 Aug;14(3):181-7. doi: 10.1111/j.1442-9071.1986.tb00034.x. PMID 3768171
- [Derived] Sen HN, Larson TA, Meleth AD, Smith WM, Nussenblatt RB. Subconjunctival sirolimus for the treatment of chronic active anterior uveitis: results of a pilot trial. Am J Ophthalmol. 2012 Jun;153(6):1038-42. doi: 10.1016/j.ajo.2011.12.018. Epub 2012 Apr 1. PMID 22465364